CLINICAL TRIAL: NCT06973928
Title: Is Change in Mouth Opening Related to Change in Quality of Life in Children With Type 1 Obstructive Sleep Apnea After Adenotonsillectomy? The JawChild Prospective Cohort Study
Brief Title: Is Change in Mouth Opening Related to Change in Quality of Life in Children With Type 1 Obstructive Sleep Apnea After Adenotonsillectomy?
Acronym: JawChild
Status: Not yet recruiting | Type: Observational
Sponsor: Groupe Adène (Other)
Collaborators: Clinique Saint Jean, France (Other); Institute of Neurosciences of Montpellier, INSERM U583 (Unknown); UMR UA11INSERM-UMIDESP Institut Desbrest d'Épidémiologie et de Santé Publique (Unknown); Service d'Information Médicale, Épidémiologie et Données de Santé (SIMED), CHU Montpellier (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024-A02761-46
Record Dates: First submitted 2025-04-04; First posted 2025-05-15 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Sleep Apnea, Obstructive
Keywords: type 1 obstructive sleep apnea; adenotonsillectomy; mouth opening; Polysomnography
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All study participants: This study is a non-randomized, monocentric, prospective trial with a non-blinded single arm. All participants need to have received a surgical indication for adenotonsillectomy to be included in the study. The participants will undergo polysomnography coupled with measurements of mouth opening (using the Jawac) before and after the adenotonsillectomy. Each participant's parent or legal guardian will also complete questionnaires that will provide information about the participant's quality of life and symptoms.
  Interventions: Device: Measures of jaw activity using the Jawac

INTERVENTIONS:
Device: Measures of jaw activity using the Jawac — At the inclusion visit (V1), informed consent will be obtained from one parent or legal guardian of each participant, who will then complete questionnaires about their children's quality of life and sleep-related symptoms. Participating children will undergo PSG combined with Jawac measurements of jaw activity. Patients will undergo adenotonsillectomy during the surgical visit (V2). Three months later, at the follow-up visit (V3), patients will again undergo PSG with Jawac measurements, and the same parent or legal guardian will complete the same questionnaires.

SUMMARY:
The goal of this clinical trial is to learn if changes in quality of life are linked to changes in mouth opening after adenotonsillectomy in a group of children who were diagnosed with Type 1 Obstructive Sleep Apnea (OSA1). The main questions it aims to answer are:

Primary Objective:

•Are changes in quality of life linked to improvements in mouth opening after adenotonsillectomy?

Secondary Objectives:

* How does quality of life change after adenotonsillectomy, based on different questionnaires about the child's sleep, breathing, behavior, and emotions?
* Is there a link between changes in quality of life and changes in mouth movements after adenotonsillectomy?
* Is there a link between changes in quality of life and changes in sleep quality after adenotonsillectomy?
* How do clinical symptoms change after adenotonsillectomy?
* Are measures of mouth movements linked to measurements of sleep quality after adenotonsillectomy?

Participation will require:

* Participating children will have adenotonsillectomy surgery, as suggested by their doctor
* Before and after tonsillectomy, parents of participating children will answer questionnaires related to their child's quality of life and their child's symptoms related to sleep, breathing, behavior, and emotions
* Sleep quality and mouth opening will be evaluated in participating children before and after tonsillectomy

DETAILED DESCRIPTION:
STUDY BACKGROUND AND OBJECTIVES Obstructive Sleep Disordered Breathing (oSDB) encompasses a range of abnormal breathing patterns during sleep, from snoring to complete airway obstruction, caused by increased upper airway resistance and pharyngeal collapsibility. Although often considered an adult disease, oSDB also occurs in children, and has been linked to metabolic, cardiovascular, and neurocognitive morbidity, and lower quality of life in pediatric patients. This study focuses on children who have Type 1 Obstructive Sleep Apnea (OSA1), a condition where a person's airway can become blocked repeatedly during sleep. The common treatment for OSA1 is adenotonsillectomy.

OSA1 is diagnosed and evaluated using the Apnea-Hypopnea Index (AHI), which is considered an indicator of OSA severity. Polysomnography (PSG), the gold standard for measuring AHI, is a time consuming and costly procedure that is impractical for follow-up in a pediatric population. Furthermore, AHI has not been shown to be related to quality of life in children with OSA1. For this reason, interest in using measuring mouth opening, instead of PSG, to evaluate OSA1 has grown. Mouth opening reflects mouth breathing, a common clinical feature of OSA1 that is linked to respiratory effort. In children with OSA1, improvements in mouth breathing have been associated with better behavior, decreased sleepiness, and increased quality of life.

The Jawac© is a novel technology that can be used to reliably measure jaw activity, which is used to evaluate mouth opening, in children. Previous research has shown that changes in respiratory effort-related arousal after adenotonsillectomy were related to changes in mandibular movement. However, no previous research has identified a straightforward, objective biomarker that correlates with quality of life and surgical outcomes in children undergoing adenotonsillectomy. Given the observed links between mouth opening, respiratory effort, and quality of life in pediatric patients, the primary objective of this clinical trial is to determine if changes in quality of life are linked to changes in mouth opening after adenotonsillectomy in a group of children who were diagnosed with OSA1. The secondary aims include studying the relationships between change in quality of life and changes in common Jawac and PSG metrics as well as evaluating variations in quality of life, changes in clinical symptoms, and the relationship between Jawac and PSG metrics in the same population of children who undergo adenotonsillectomy.

STUDY DESIGN AND METHODS This research study is non-randomized, monocentric, prospective, and features a single non-blinded arm due to its exploratory and descriptive nature. During the pre-inclusion visit (V0), surgeons will screen patients for eligibility to participate in the study. At the inclusion visit (V1), informed consent will be obtained from one parent or legal guardian of each participant, who will then complete questionnaires about their children's quality of life and sleep-related symptoms. Participating children will undergo PSG combined with Jawac measurements. The adenotonsillectomy will occur during the surgical visit (V2). Three months later, at the follow-up visit (V3), patients will again undergo PSG with Jawac measurements, and the same parent or legal guardian will complete the same questionnaires. Four months post-surgery, patients will have a follow-up consultation with the surgeon (V4). The study protocol adheres to national guidelines for standard OSA management, with the addition of the questionnaires at V1 and V3, and the PSG with Jaw activity (measured using the Jawac) measurement at V3. Only one extra consultation (V3) is added to the standard patient pathway, thus a low rate of study discontinuation is anticipated. Data from patients who discontinue or deviate from the intervention will be excluded. Adverse events will be documented throughout the study at V1, V2, V3, and V4.

ELIGIBILITY:
Inclusion Criteria:

* Age: 3 to 7 years old
* Received a surgical indication for adenotonsillectomy
* Beneficiary of the French single-payer national medical insurance system
* Informed consent given
* Able to attend all scheduled visits and comply with all trial procedures.

Exclusion Criteria:

* Previous adenotonsillectomy
* Subject has already participated in the current study
* Craniofacial malformation syndrome
* BMI according to age > 97th percentile
* Previous or current stimulant medication (methylphenidate)
* Current orthodontic treatment
* Asymmetric score of the tonsil with a tonsil Brodsky score of ≤2
* Subject who are in a dependency or employment with the sponsor or the investigator
* Participation in another clinical trial or administration of an unapproved drug within the last 4 weeks before the screening date

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will include pediatric patients between the ages of three and seven years old, who consulted with a surgeon at the study center for potential adenotonsillectomy. To be eligible to participate, patients must be beneficiaries of the French single payer national medical insurance system, be able to attend all scheduled visits and comply with trial procedures, and legal guardians must give informed consent. Full inclusion and exclusion criteria are listed in Table 1. The study center is a private French hospital that, due to the single-payer insurance system in France, should include patients from a range of socioeconomic categories and geographical (urban versus rural) locations.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Correlation between change in quality of life and change in mouth opening | Change from the inclusion visit (V1) to three months after adenotonsillectomy (V3).
  Quality of life (QOL) will be evaluated using two versions of the Pediatric Quality of Life Inventory Parent Proxy Report (PedsQL PPR). The PedsQL PPR 2-4 will be used for participants 3-4 years old, and the PedsQL PPR 5-7 will be used for participants 5-7 years old. For both versions, total scores range from 0-100 points. Higher scores indicate better health related QOL.
  The JAWAC sensor will be used to measure Mouth Opening in 1/10 millimeters to assess oral breathing during sleep. Oral breathing is a potential cause of sleep apnea in children. Higher measures of Mouth Opening (in millimeters) indicates a greater degree of respiratory disturbance during sleep.
  The main endpoint analysis (correlation between change in QOL and change in Mouth Opening) will be done using the estimation of the ρ coefficient. A linear regression will be used for the analysis before and after adjustment for confounding variables.

SECONDARY OUTCOMES:
Changes in quality of life | Change from the inclusion visit (V1) to three months after adenotonsillectomy (V3).
  QOL will be evaluated using two versions of the Pediatric Quality of Life Inventory Parent Proxy Report (PedsQL PPR). The PedsQL PPR 2-4 will be used for participants 3-4 years old, and the PedsQL PPR 5-7 will be used for participants 5-7 years old. For both versions, total scores range from 0-100 points. Higher scores indicate better health related QOL.
  The same parent or legal guardian will complete the PedsQL at inclusion (V1) and three months after adenotonsillectomy (V3)
The correlations between changes in quality of life and changes in other mandibular movement metrics | Change from the inclusion visit (V1) to three months after adenotonsillectomy (V3).
  Quality of life (QOL) will be evaluated using two versions of the Pediatric Quality of Life Inventory Parent Proxy Report (PedsQL PPR). The PedsQL PPR 2-4 will be used for participants 3-4 years old, and the PedsQL PPR 5-7 will be used for participants 5-7 years old. For both versions, total scores range from 0-100 points. Higher scores indicate better health related QOL.
  The mandibular movement (MM) measures that will be evaluated using the Jawac are: large MM (MML): the number of MM amplitudes ≥0.3 mm from peak to peak during ≥two respiratory cycles; Sharp MM (MMS): the number of sudden large MMs (amplitude >1mm and/or amplitude ≥200% of the previous and/or the ensuing MM amplitude) during one respiratory cycle; Mandibular movement opening (MMO): how wide the mouth opens (in mm) during MM; Time durations during non-rapid eye movement sleep when mandibular movement is higher than 0.4 mm (tMM0.4), 0.3 mm (tMM0.3), and 0.2 mm (tMM0.2).
  Correlation analyses will be conducted
The relationship between changes in quality of life and changes in polysomnography respiratory disturbance index | Change from the inclusion visit (V1) to three months after adenotonsillectomy (V3).
  Quality of life (QOL) will be evaluated using two versions of the Pediatric Quality of Life Inventory Parent Proxy Report (PedsQL PPR). The PedsQL PPR 2-4 will be used for participants 3-4 years old, and the PedsQL PPR 5-7 will be used for participants 5-7 years old. For both versions, total scores range from 0-100 points. Higher scores indicate better health related QOL.
  Polysomnography respiratory disturbance index (PSG-RDI), which measures the number of abnormal breathing events per hour of sleep, will be evaluated as defined by the American Academy of Sleep Medicine 2018. PSG-RDI defines sleep apnea severity as follows: normal: <5 events/hr; mild: ≥5 but <15 events/hr; moderate: ≥15 but <30 events/hr; severe: ≥30 events/hr.
  A linear regression will be used for the analysis before and after adjustment for confounding variables
Changes in the Sleep-related Breathing Disorder scale | Change from the inclusion visit (V1) to three months after adenotonsillectomy (V3).
  Clinical symptoms will be evaluated using The Sleep-related Breathing Disorder scale of the Pediatric Sleep Questionnaire (PSQ), which consists of 22 items. The score is the mean response on non-missing items, which can vary from 0 to 1. Higher scores reflect high risk for a pediatric sleep-related breathing disorder.
Correlations between mandibular movement and Polysomnography respiratory disturbance index | Change from the inclusion visit (V1) to three months after adenotonsillectomy (V3).
  The mandibular movement (MM) measures that will be evaluated using the Jawac are: large MM (MML): the number of MM amplitudes ≥0.3 mm from peak to peak during ≥two respiratory cycles; Sharp MM (MMS): the number of sudden large MMs (amplitude >1mm and/or amplitude ≥200% of the previous and/or the ensuing MM amplitude) during one respiratory cycle; Mandibular movement opening (MMO): how wide the mouth opens (in mm) during MM; Time durations during non-rapid eye movement sleep when mandibular movement is higher than 0.4 mm (tMM0.4), 0.3 mm (tMM0.3), and 0.2 mm (tMM0.2).
  Polysomnography respiratory disturbance index (PSG-RDI), which measures the number of abnormal breathing events per hour of sleep, will be evaluated as defined by the American Academy of Sleep Medicine 2018. PSG-RDI defines sleep apnea severity as follows: normal: <5 events/hr; mild: ≥5 but <15 events/hr; moderate: ≥15 but <30 events/hr; severe: ≥30 events/hr.
  Correlation analyses will be conducted
Changes in acute sleep disturbances | Change from the inclusion visit (V1) to three months after adenotonsillectomy (V3)
  The Sleep Disturbance Scale for Children (SDSC) (separate versions for 3-4 and for 5-7 year olds) has 26 items, scored from 1-5 (maximmum score 130, minimum score 1). Higher scores indicate more acute sleep disturbances.
Changes in emotional and behavioral difficulties | Change from the inclusion visit (V1) to three months after adenotonsillectomy (V3)
  The Strengths and Difficulties Questionnaire (SDQ) (separate versions for 3-4 and 5-7 year olds) has 25 items divided into 5 scales (score range: 0-40). Higher total scores suggest significant emotional and behavioral difficulties.
Severity Hierarchy Score for Respiratory Symptoms | Change from the inclusion visit (V1) to three months after adenotonsillectomy (V3)
  The Severity Hierarchy Score (SHS) will be used to rank respiratory symptoms from least to most severe. It does not have defined maximum and minimum scores.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Akkari, MD, Principal Investigator — Clinique Saint Jean, France
Locations (1):
- Clinique Saint Jean, Saint-Jean-de-Védas, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goodman R. The Strengths and Difficulties Questionnaire: a research note. J Child Psychol Psychiatry. 1997 Jul;38(5):581-6. doi: 10.1111/j.1469-7610.1997.tb01545.x. PMID 9255702
- [Background] Bruni O, Ottaviano S, Guidetti V, Romoli M, Innocenzi M, Cortesi F, Giannotti F. The Sleep Disturbance Scale for Children (SDSC). Construction and validation of an instrument to evaluate sleep disturbances in childhood and adolescence. J Sleep Res. 1996 Dec;5(4):251-61. doi: 10.1111/j.1365-2869.1996.00251.x. PMID 9065877
- [Background] Rosen CL, Wang R, Taylor HG, Marcus CL, Katz ES, Paruthi S, Arens R, Muzumdar H, Garetz SL, Mitchell RB, Jones D, Weng J, Ellenberg S, Redline S, Chervin RD. Utility of symptoms to predict treatment outcomes in obstructive sleep apnea syndrome. Pediatrics. 2015 Mar;135(3):e662-71. doi: 10.1542/peds.2014-3099. Epub 2015 Feb 9. PMID 25667240
- [Background] Jordan L, Beydon N, Razanamihaja N, Garrec P, Carra MC, Fournier BP, Vi-Fane B, Kerner S, Felizardo R, Boy-Lefevre ML, De La Dure-Molla M. Translation and cross-cultural validation of the French version of the Sleep-Related Breathing Disorder scale of the Pediatric Sleep Questionnaire. Sleep Med. 2019 Jun;58:123-129. doi: 10.1016/j.sleep.2019.02.021. Epub 2019 Mar 14. PMID 31146124
- [Background] Chervin RD, Hedger K, Dillon JE, Pituch KJ. Pediatric sleep questionnaire (PSQ): validity and reliability of scales for sleep-disordered breathing, snoring, sleepiness, and behavioral problems. Sleep Med. 2000 Feb 1;1(1):21-32. doi: 10.1016/s1389-9457(99)00009-x. PMID 10733617
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Aubertin G, Akkari M, Andrieux A, Colas des Francs C, Fauroux B, Franco P, Gagnadoux F, de Santerre OG, Grollemund B, Hartley S, Jaffuel D, Lafond L, Schroder CM, Schweitzer C, Charley-Monaca C. Management of obstructive sleep apnea syndrome type 1 in children and adolescents - A French consensus. Arch Pediatr. 2023 Oct;30(7):510-516. doi: 10.1016/j.arcped.2023.06.009. Epub 2023 Aug 2. PMID 37537084
- [Background] Costain G, Cohn RD, Malkin D. Precision Child Health: an Emerging Paradigm for Paediatric Quality and Safety. Curr Treat Options Pediatr. 2020;6(4):317-324. doi: 10.1007/s40746-020-00207-2. Epub 2020 Aug 25. PMID 38624480
- [Background] Martinot JB, Le-Dong NN, Denison S, Guenard HJ, Borel JC, Silkoff PE, Pepin JL, Gozal D. Persistent respiratory effort after adenotonsillectomy in children with sleep-disordered breathing. Laryngoscope. 2018 May;128(5):1230-1237. doi: 10.1002/lary.26830. Epub 2017 Aug 22. PMID 28833232
- [Background] Bandyopadhyay A, Slaven JE. Health outcomes associated with improvement in mouth breathing in children with OSA. Sleep Breath. 2021 Sep;25(3):1635-1639. doi: 10.1007/s11325-020-02247-2. Epub 2021 Jan 7. PMID 33411187
- [Background] Leal RB, Gomes MC, Granville-Garcia AF, Goes PS, de Menezes VA. Impact of breathing patterns on the quality of life of 9- to 10-year-old schoolchildren. Am J Rhinol Allergy. 2016 Sep;30(5):147-52. doi: 10.2500/ajra.2016.30.4363. PMID 27657891
- [Background] Liu X, Immanuel S, Pamula Y, Kennedy D, Martin J, Baumert M. Adenotonsillectomy for childhood obstructive sleep apnoea reduces thoraco-abdominal asynchrony but spontaneous apnoea-hypopnoea index normalisation does not. Eur Respir J. 2017 Jan 25;49(1):1601177. doi: 10.1183/13993003.01177-2016. Print 2017 Jan. PMID 27811072
- [Background] Mitchell RB, Garetz S, Moore RH, Rosen CL, Marcus CL, Katz ES, Arens R, Chervin RD, Paruthi S, Amin R, Elden L, Ellenberg SS, Redline S. The use of clinical parameters to predict obstructive sleep apnea syndrome severity in children: the Childhood Adenotonsillectomy (CHAT) study randomized clinical trial. JAMA Otolaryngol Head Neck Surg. 2015 Feb;141(2):130-6. doi: 10.1001/jamaoto.2014.3049. PMID 25474490
- [Background] da Silva Gusmao Cardoso T, Pompeia S, Miranda MC. Cognitive and behavioral effects of obstructive sleep apnea syndrome in children: a systematic literature review. Sleep Med. 2018 Jun;46:46-55. doi: 10.1016/j.sleep.2017.12.020. Epub 2018 Feb 9. PMID 29773210
- [Background] Katz ES, D'Ambrosio CM. Pathophysiology of pediatric obstructive sleep apnea. Proc Am Thorac Soc. 2008 Feb 15;5(2):253-62. doi: 10.1513/pats.200707-111MG. PMID 18250219
- [Derived] Akkari M, Lopez R, Jaussent I, Vidal C, Skinner S, Jaffuel D, Molinari N. Is a change in mouth opening associated with improvements in quality of life in children with type 1 obstructive sleep apnoea after adenotonsillectomy? Protocol for the JawChild prospective cohort study. BMJ Open. 2025 Dec 14;15(12):e105324. doi: 10.1136/bmjopen-2025-105324. PMID 41397757